CLINICAL TRIAL: NCT04796402
Title: A Pragmatic Eight Week Phase IV Study of Bamlanivimab/LY-CoV555 for Emergency Passive Immunity Against COVID-19
Brief Title: A Study to Assess if a Medicine Called Bamlanivimab is Safe and Effective in Reducing Hospitalization Due to COVID-19
Acronym: B-EPIC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fraser Health (Other)
Collaborators: Fraser Health Authrority Department of Evaluation and Research Services (Unknown); Surrey Memorial Hospital Clinical Research Unit (Unknown); Centre for Health Evaluation and Outcome Sciences (Unknown); Surrey Hospital Foundation (Unknown); BC Support Unit (Other); University of British Columbia (Other); Ministry of Health, British Columbia (Other Government); Clinical Trials BC (part of the BC Academic Health Science Network) (Unknown)
Responsible Party: Principal Investigator, Gregory Haljan, MD, Principal Investigator, Fraser Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FHREB 2021-023
Record Dates: First submitted 2021-03-10; First posted 2021-03-12 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Covid19
Keywords: Bamlanivimab; monoclonal antibody; hospitalization; mortality; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — bamlanivimab; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control (Active Comparator): Standard of care
  Interventions: Other: Standard of Care
- Intervention (Experimental): Administration of Bamlanivimab
  Interventions: Biological: Bamlanivimab

INTERVENTIONS:
Biological: Bamlanivimab — 700 mg/20mL IV over at least one hour OD
  Arms: Intervention
Other: Standard of Care — Standard of care includes primary care and specialist care as indicated by the patient's primary care provider
  Arms: Control

SUMMARY:
The purpose of this research is to test whether a new medication called bamlanivimab is safe and effective at reducing the need for hospitalization due to COVID-19.

DETAILED DESCRIPTION:
The study aims to examine the effectiveness of adding bamlanivimab provided by COVID-19 Clinics to standard of care on the incidence of hospitalization for high-risk patients infected with SARS-CoV2. Furthermore, we aim to test the effect on the following secondary outcomes: mortality and health-related quality of life and patients' satisfaction with care. We will also assess the recruitment rate from the three primary strategies for rapid identification and consent of eligible patients. The data from this study will inform clinical decisions about the use of bamlanivimab in high risk COVID-19 patients and the operational requirements necessary for research in passive immunity therapeutics.

ELIGIBILITY:
Inclusion Criteria:

1. Age at the time of SARS-CoV2 test:

   1. Age > 65
   2. Age 55-64 and 1 or more of:

   i. BMI>35, ii. chronic kidney disease, iii. diabetes mellitus, iv. immunosuppressive disease v. current immunosuppressive treatment vi. hypertension vii. coronary artery disease viii. chronic lung disease

   c. Age 18-54 and 1 or more of: i. BMI>35 ii. chronic kidney disease iii. diabetes mellitus iv. immunosuppressive disease v. current immunosuppressive treatment
2. Disease Characteristics:

   1. Not hospitalized
   2. Sample collection for first SARS-CoV2 test positive within 3 days prior to consent.
   3. One or more mild COVID-19 symptoms and within 10 days from onset

   i. Fever ii. Cough iii. Sore throat iv. Malaise v. Headache vi. Muscle pain vii. Gastrointestinal symptoms viii. Shortness of breath with/without exertion
3. Study Procedures:

   1. Resident of British Columbia
   2. Understand and agree to planned study procedures
4. Ability and Willingness to Provide Informed Consent:

The participant will provide informed consent by telephone

Exclusion Criteria:

1. Medical Conditions

   1. Allergies to any of the components used in the formulation of the bamlanivimab
   2. Hospitalization or expected to need hospitalization in the next 24 hours at the time of recruitment for COVID-19
   3. Suspected or proven infection other than COVID-19 that in the opinion of the clinicians could pose a risk to study inclusion
   4. Any co-morbidity considered life-threatening in <28 days, or requiring surgery in <7 days.
   5. Any serious disease, condition or disorder that in the opinion of the clinicians should preclude participation.
   6. Require oxygen therapy due to COVID-19
   7. Require an increase in baseline oxygen flow rate due to COVID-19 in those on chronic oxygen therapy due to underlying non-COVID-19 related comorbidity.
2. Weighs < 40 kg
3. History of vaccination against SARS-CoV2
4. History of convalescent plasma or IVIG therapy within 3 months of first SARS-CoV2 viral determination positive
5. History of previous SARS-CoV2 infection
6. History of participation in any clinical study involving an investigational intervention within 30 days or 5 half-lives of the previous intervention, whichever is longer.
7. Unable to achieve informed consent for any reason
8. Known Pregnancy
9. Actively breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 576 (Estimated)
Dates: Start 2021-03-17 (Actual); Primary Completion 2021-06-07 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Any incidence of admission to hospital for >24 hours in the 28 days following first positive test for SARS-CoV2. | 0 - 28 days following first positive test for COVID 19

SECONDARY OUTCOMES:
Any incidence of admission to hospital for >24 hours following first positive test for SARS-CoV2. | 0 - 28 days following first positive test for COVID-19
Mortality following first positive test for SARS-CoV2. | 28 days, 3 month and 6 months post-treatment
Health-related quality of life assessment. | Screening and 6 months post-treatment
  Medical Outcomes Study: 20-Item Short Form Survey Instrument (SF-20)
Hospitalization by age and comorbidities. | Treatment day and up to 6 months post-treatment
Incidence and types of adverse reactions including anaphylaxis. | Treatment day and up to 6 months post-treatment
Recruitment rate. | Upto 8 weeks from day of first patient recruited to day of last patient recruited
Overall satisfaction with participation in research. | 6 months post-treatment
  Likert Scale
Type and frequency of viral variants in patients receiving bamlanivimab. | Up to 8 weeks from day of first patient recruited to day of last patient recruited

CONTACTS AND LOCATIONS:
Locations (1):
- Fraser Health Authority, Fraser Health Region, British Columbia, Canada

REFERENCES:
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343